CLINICAL TRIAL: NCT03473990
Title: A Randomised Control Trial to Assess the Efficacy of Short-term, Home-based High- Intensity Interval Training (HIT) for Improving Indices of Cardiorespiratory Fitness
Brief Title: Short-term, Home-based, High-intensity Interval Training (HIT) for Improving Fitness
Acronym: HomeHIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Bethan Phillips, Assistant Professor, University of Nottingham
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: C16122016
Record Dates: First submitted 2017-10-31; First posted 2018-03-22 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: High-Intensity Interval Training
Keywords: Home-based; Short-term; Randomised Control Trial
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laboratory HIT (Active Comparator): Supervised (Laboratory HIT) exercise in the lab up to 4 times per week for 4 weeks
  Interventions: Other: High-intensity interval training
- Home HIT (Active Comparator): Unsupervised (Home HIT) exercise at home up to 4 times per week for 4 weeks
  Interventions: Other: High-intensity interval training
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Other: High-intensity interval training — 2 minute warm up, followed by 5x1min HIT intervals separated by 90 seconds active recovery (walking on the spot) and then a 2 minute recovery period. The high intensity bouts will be a pyramid of exercises (star jumps, mountain climbers and on-the-spot sprints)
  Other Names: HIT
  Arms: Home HIT; Laboratory HIT

SUMMARY:
This study will aim to evaluate the efficacy of a short-term, home-based, high-intensity interval (HIT) programme in improving cardiovascular fitness in healthy volunteers aged 55 and above, with an age-comparison to younger individuals taking part in the same training regime.

It will also explore the efficacy of time-matched 'static' interventions for improving cardiovascular parameters in middle-aged females and older adults.

DETAILED DESCRIPTION:
Patients with lower peak oxygen uptake have higher mortality and morbidity when undergoing major surgery. Aerobic fitness is a potentially modifiable risk factor for postoperative complications.

Traditional pre-operative exercise interventions to improve fitness involve high time and supervision-demands, often resulting in poor compliance. High-intensity interval training (HIT) is a time-efficient, feasible method to improve pre-operative fitness, however current studies only involve exercise in the laboratory setting.

Study Design Thirty-six healthy volunteers aged 55y and over will be randomly allocated to one of three groups: 1) Laboratory-HIT; 2) Home-HIT; 3) No intervention. All HIT sessions will involve a brief warm-up, followed by five 1-minute bouts of high-intensity (body-weight based) exercise, interspersed with 90-seconds recovery, concluding with a brief cool-down. The primary endpoint of the study is change in VO2 peak with secondary endpoints of changes in: anaerobic threshold, insulin sensitivity and muscle mass.

Subjects will be expected to perform up to a maximum of 16 HIT sessions (maximum 5 sessions per week) within a period of 31 days. Aerobic fitness will be assessed prior to and following the exercise, as will body composition, muscle structure, physical function and insulin sensitivity.

For the age comparison, 24 young individuals will be recruited to either a control or home-HIT arm.

In addition, the efficacy of time-matched 'static' interventions for improving cardiovascular parameters in 24 middle-aged females will also be assessed as exploratory work for these interventions.

The efficacy of the static interventions in older adults at home will also be explored.

Power calculation: The investigators performed a power calculation for the primary outcome of VO2 max in older adults using data from a previous study at our centre on home versus laboratory HIIT. Assuming an effect size F of 0.6 for three groups and a within group SD of 5, the alpha level was set at 0.05 and the 1-beta at 0.80. This concluded that 30 participants would be required. To allow for potential non-completion and missing data 36 older participants will be enrolled to the study (12 to each group).

ELIGIBILITY:
Inclusion Criteria:

Age > 55 years Able to give informed consent

Exclusion Criteria:

* Current participation in a formal exercise regime
* A BMI < 18 or > 35 kg·m2
* Active cardiovascular disease:

  * Uncontrolled hypertension (BP > 160/100)
  * Angina
  * Heart failure (class III/IV)
  * Significant arrhythmia
  * Right to left cardiac shunt
  * Recent cardiac event
* Taking beta-adrenergic blocking agents
* Cerebrovascular disease:

  * Previous stroke
  * Aneurysm (large vessel or intracranial)
  * Epilepsy
* Respiratory disease including:

  * Pulmonary hypertension
  * Significant COPD
  * Uncontrolled asthma
* Malignancy
* Metabolic disease e.g. diabetic patients
* Clotting dysfunction
* Significant Musculoskeletal or neurological disorders
* Family history of early (<55y) death from cardiovascular disease

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Change in VO2 Max (L/min) assessed by Cardio-pulmonary exercise test (CPET) | 31 days
  To determine the efficacy of bodyweight HIT for improving aerobic fitness

SECONDARY OUTCOMES:
Change in Anaerobic Threshold (L/min) using CPET | 31 days
  To determine the efficacy of bodyweight HIT for improving aerobic fitness
Change in resting glucose and insulin sensitivity (mmol/L) | 31 days
  The effects of HIT on improving glucose control using Oral Glucose Tolerance Test (OGTT) and enzyme-linked immunosorbent assay (ELISA)
Change in muscle architecture as assessed by ultrasound | 31 days
  To assess the effects of HIT on improving muscle structure and function
Change in body composition (fat, muscle, bone (g)) as assessed by Dual-energy Xray Absorptiometry (DEXA) | 31 days
  To assess the effects of HIT on improving muscle structure and function
Feasibility of home HIT assessed using a preset feasibility questionnaire | 31 days
  To assess the feasibility and acceptability of performing a HIT programme at home

CONTACTS AND LOCATIONS:
Overall Officials: Bethan Philips, Principal Investigator — The University of Nottingham, Division of Medical Sciences and Graduate Entry Medicine, School of Medicine, Royal Derby Hospital, Derby, DE22 3DT
Locations (1):
- The University of Nottingham, Division of Medical Sciences and Graduate Entry Medicine, School of Medicine, Royal Derby Hospital, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable participant data will be made available for all outcome measures
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Duration of PhD (3 years)
Access Criteria: Password protected database only given to researchers with special access to the database

REFERENCES:
- [Derived] Sian TS, Inns TB, Gates A, Doleman B, Bass JJ, Atherton PJ, Lund JN, Phillips BE. Equipment-free, unsupervised high intensity interval training elicits significant improvements in the physiological resilience of older adults. BMC Geriatr. 2022 Jun 28;22(1):529. doi: 10.1186/s12877-022-03208-y. PMID 35761262